CLINICAL TRIAL: NCT03156660
Title: Efficacy of Two Novel Behavioral Post-cessation Weight Gain Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Mayo Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-04522-FB; R01DK107747 (NIH)
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-04

CONDITIONS: Weight Change, Body; Smoking Cessation
MeSH Terms: conditions — Body Weight Changes; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight gain prevention (Group 1) (Experimental): Small Changes weight stability intervention
  Interventions: Behavioral: Weight gain prevention (Group 1)
- Weight loss intervention (Group 2) (Experimental): Look AHEAD weight loss intervention
  Interventions: Behavioral: Weight loss intervention (Group 2)
- Self-guided intervention (Group 3) (Active Comparator): Self-guided weight management with the EatingWell Diet book
  Interventions: Behavioral: Self-guided intervention (Group 3)

INTERVENTIONS:
Behavioral: Weight gain prevention (Group 1) — Participants will be asked to keep their weight stable during the initial 8 weeks of the study.
  Intervention Components:
  1. Lesson materials adapted from the Small Changes intervention, which will provide guidance for meeting the goals of this intervention (i.e., increasing steps by 2000 steps per day, making one Small dietary Change each day).
  2. Daily self-monitoring of steps and number of Small Changes
  3. Daily weight self-monitoring on the BodyTraceTM e-scale
  4. Fit Bit Alta activity trackers to self-monitor steps
  Arms: Weight gain prevention (Group 1)
Behavioral: Weight loss intervention (Group 2) — Participants will be asked to achieve a weight loss goal of at least 5% of their baseline weight by week 8.
  Intervention Components:
  1. Tailored calorie and fat goals based on their baseline weight.
  2. Daily dietary intake and physical activity self-monitoring using a website or app.
  3. Daily weight self-monitoring on the BodyTraceTM e-scale
  4. Lesson materials for each session, drawn from the Look AHEAD intensive lifestyle intervention
  5. Meal replacements for two meals and one snack for 8 weeks as a method to achieve the study's calorie and fat goals and as a strategy to control portions
  6. Graded physical activity goals of 175 minutes of moderate intensity exercise (e.g., brisk walking) per week, or 10,000 steps per day
  7. Fit Bit Alta activity trackers to self-monitor steps
  Arms: Weight loss intervention (Group 2)
Behavioral: Self-guided intervention (Group 3) — Participants randomized to Group 3 will wait for 8 weeks before initiating the same smoking cessation intervention as the other two conditions, while they review the provided weight management focused book.
  Intervention Components:
  1. EatingWell Diet book.
  2. Daily weight self-monitoring on the BodyTraceTM e-scale
  Arms: Self-guided intervention (Group 3)

SUMMARY:
The study aims to randomize 400 participants to 1 of 3 arms: a) a weight stability intervention prior to smoking cessation (Group 1); b) a weight loss intervention prior to smoking cessation (Group 2); or c) a self-guided weight management prior to cessation (Group 3) and to determine the efficacy of the interventions on preventing weight gain at 12 month follow-up. All 3 conditions receive a highly efficacious behavioral smoking cessation program and 6 months of varenicline pharmacotherapy (ChantixTM), the most efficacious medication for smoking cessation.

DETAILED DESCRIPTION:
While smoking cessation leads to significant improvements in mortality and morbidity, weight gain post-cessation partially attenuates this benefit. Furthermore, concerns about postcessation weight gain are common and are often cited as a reason to delay cessation attempts. In addition, postcessation weight gain is associated with smoking relapse. Thus, although the health benefits of smoking cessation outweigh the negative impact of weight gain, ideally there would be intervention "packages" that would not require that people choose between smoking cessation and nontrivial weight gain. Thus, in the proposed study, the investigators will determine whether two very promising methods of reducing postcessation weight gain, namely a weight stability intervention (based on the evidence-based Small Changes intervention) versus a weight loss intervention (based on the evidence-based Look AHEAD intensive lifestyle intervention) followed by a smoking cessation intervention are efficacious for reducing postcessation weight gain. The investigators will randomize 400 smokers to one of three arms: a) a weight stability intervention prior to cessation (Group 1); b) a weight loss intervention prior to cessation (Group 2), or c) a self-guided intervention prior to cessation (Group 3) and to determine the efficacy of the interventions on preventing weight gain at 12 month follow-up. All three conditions receive a highly efficacious in-person smoking cessation behavioral intervention and six months of Varenicline (ChantixTM) pharmacotherapy. Those participants randomized to the Group 1 and Group 2 conditions will receive monthly booster weight management sessions, after completing the behavioral smoking cessation intervention. The primary outcomes will be weight change and smoking cessation at 12 month follow-up. In addition, the investigators will gather process data on mediators of treatment outcome via measures of treatment engagement (e.g., session attendance, varenicline utilization). The investigators will be able to determine whether a weight stability intervention or a weight loss intervention is efficacious in reducing post-cessation weight gain. The intervention results, if successful, could be disseminated and make a significant contribution towards curtailing obesity in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Participants must wish to quit smoking in the next 30 days
* Have smoked 5 or more cigarettes a day for at least 1 year
* Participants must be 18 years or older as the safety and efficacy of varenicline therapy has not been established for pediatric patients
* Participants must have a BMI of 22 kg/m2 or greater, as it would not be recommended to have those who are underweight or the lower end of the normal BMI range attempt a 5% weight loss (if assigned to the Group 2 condition)
* Participants must have access to a telephone and daily access to email, if using a cell phone, participants must be willing to use their cell phone minutes for weekly phone interventions
* Participants must have the ability to understand consent process in English
* If female and of childbearing age, participant must have a negative pregnancy test and must agree to use contraception during participation in the study
* All participants must be willing to be randomized to the study conditions and wait eight weeks prior to beginning smoking cessation (during which they will participate in the weight management intervention to which they are assigned).
* Participants must have BP < 150/95 and a heart rate of >40 beats per minute and <120 beats per minute.

Exclusion Criteria:

* Participants must not have a known contraindication, allergy or hypersensitivity to varenicline therapy
* Participants must not currently (in the previous 30 days) be participating in other behavioral or pharmacologic weight or smoking cessation interventions
* Participants must not have had weight loss surgery (hx of gastric bypass, stomach stapling or banding)
* Participants must not have lost > or equal to10 lbs in the past 6 months
* Participants must not be taking a medication that impacts weight
* Participants must not have used an investigational drug within the last 30 days
* Participants must not have current suicidal thoughts or have a lifetime history of a suicide attempt as defined by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Participants must not self-report a history of psychosis, bipolar disorder, or anorexia nervosa
* Participants must not have self-reported current alcohol abuse or illicit substance use
* Participants must not have kidney or liver disease, unstable cardiovascular conditions, HIV, or history of cancer in last 5 years
* Participants must not have another member of their household already participating in this study
* Participants must not be currently pregnant or lactating or planning to become pregnant in the next 12 months, or have been pregnant within the last 6 months
* Weight limit of 385 pounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Krukowski, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that a cleaned data set of study-specific data will be provided within two years following the termination of the study for the data archive and this data set would be made public. Confidentiality of individual participants would be maintained with all releases of data. The final study analytical database would be processed according to HIPAA definitions for public data sharing. Documentation would be provided along with the data sharing file that includes but is not limited to: data dictionary, data code book, valid variable ranges (where provided), the protocol, procedure and operational manuals, intervention manual or programs and any electronic versions of any paper forms that were used in data collection.
Time Frame: Two years following the termination of the study
Access Criteria: Upon reasonable request to the principal investigator, Rebecca Krukowski

REFERENCES:
- [Derived] Pebley K, Bursac Z, Klesges RC, Ebbert JO, Womack CR, Graber J, Little MA, Derefinko KJ, Krukowski RA. A randomized controlled trial to reduce post-cessation weight gain. Int J Obes (Lond). 2023 Jun;47(6):471-478. doi: 10.1038/s41366-023-01286-5. Epub 2023 Feb 25. PMID 36841886
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902

RESULTS

PARTICIPANT FLOW:
Groups:
- Weight Gain Prevention (Group 1): Small Changes weight stability intervention
  Weight gain prevention (Group 1): Participants will be asked to keep their weight stable during the initial 8 weeks of the study.
  Intervention Components:
  1. Lesson materials adapted from the Small Changes intervention, which will provide guidance for meeting the goals of this intervention (i.e., increasing steps by 2000 steps per day, making one Small dietary Change each day).
  2. Daily self-monitoring of steps and number of Small Changes
  3. Daily weight self-monitoring on the BodyTraceTM e-scale
  4. Fit Bit Alta activity trackers to self-monitor steps
- Weight Loss Intervention (Group 2): Look AHEAD weight loss intervention
  Weight loss intervention (Group 2): Participants will be asked to achieve a weight loss goal of at least 5% of their baseline weight by week 8.
  Intervention Components:
  1. Tailored calorie and fat goals based on their baseline weight.
  2. Daily dietary intake and physical activity self-monitoring using a website or app.
  3. Daily weight self-monitoring on the BodyTraceTM e-scale
  4. Lesson materials for each session, drawn from the Look AHEAD intensive lifestyle intervention
  5. Meal replacements for two meals and one snack for 8 weeks as a method to achieve the study's calorie and fat goals and as a strategy to control portions
  6. Graded physical activity goals of 175 minutes of moderate intensity exercise (e.g., brisk walking) per week, or 10,000 steps per day
  7. Fit Bit Alta activity trackers to self-monitor steps
- Self-guided Intervention (Group 3): Self-guided weight management with the EatingWell Diet book
  Self-guided intervention (Group 3): Participants randomized to Group 3 will wait for 8 weeks before initiating the same smoking cessation intervention as the other two conditions, while they review the provided weight management focused book.
  Intervention Components:
  1. EatingWell Diet book.
  2. Daily weight self-monitoring on the BodyTraceTM e-scale
Period: Overall Study
Arm/Group | Weight Gain Prevention (Group 1) | Weight Loss Intervention (Group 2) | Self-guided Intervention (Group 3)
Started | 109 | 110 | 86
Completed | 95 | 100 | 78
Not Completed | 14 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Gain Prevention (Group 1) | Weight Loss Intervention (Group 2) | Self-guided Intervention (Group 3) | Total
Number analyzed (Participants) | 109 | 110 | 86 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (11.4) | 55.5 (11.7) | 53.8 (11.7) | 54.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 72 | 60 | 207
  Male | 34 | 38 | 26 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 4 | 6
  Not Hispanic or Latino | 107 | 110 | 82 | 299
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 50 | 46 | 36 | 132
  White | 54 | 60 | 45 | 159
  More than one race | 4 | 3 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 109 | 110 | 86 | 305
Baseline weight [Mean (Standard Deviation); unit: kilograms] — weight at baseline visit, except for 3 missing we used weight at randomization visit (occurred within 3 months from baseline visit)
  kilograms | 92.5 (21.6) | 88.2 (19.8) | 89.7 (19.9) | 90.2 (21.8)
Average number of cigarettes smoked per day [Mean (Standard Deviation); unit: number of cigarettes] — Q. 2 of Fagerstrom questionnaire at Screening Visit "How many cigarettes per day have you smoked on average in the past 7 days?"
  For out of range values, Q4 of Smoking History questionnaire at Screening Visit was used "Within the past year, how many cigarettes a day have you smoked (on average)?"
  number of cigarettes | 16.3 (8.3) | 15.9 (8.4) | 15.7 (8.8) | 15.9 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: At all measurement visits, weight will be recorded in kilograms. Weight will be measured on a calibrated digital scale in duplicate, with the participant wearing light clothing and no shoes.
Time Frame: 12 months from randomization
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Weight Gain Prevention (Group 1) | Weight Loss Intervention (Group 2) | Self-guided Intervention (Group 3)
Number analyzed (Participants) | 109 | 110 | 86
kilograms | -0.24 (0.25) | -1.11 (0.20) | 1.25 (0.27)

2. Primary Outcome: Point Prevalence Tobacco Abstinence
Description: Point prevalence (7 days without a cigarette, "not even a puff") is an appropriate measure in measuring long term outcome in cessation induction trials.
Time Frame: 12 months from randomization
Population: Completers
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Gain Prevention (Group 1) | Weight Loss Intervention (Group 2) | Self-guided Intervention (Group 3)
Number analyzed (Participants) | 95 | 100 | 80
Participants | 39 | 49 | 41

ADVERSE EVENTS:
Time Frame: 12 months
Description: Consistent with the typical definition
Arm/Group | Weight Gain Prevention (Group 1) | Weight Loss Intervention (Group 2) | Self-guided Intervention (Group 3)
All-Cause Mortality (participants affected / at risk) | 1/109 | 0/110 | 0/86
Serious Adverse Events (participants affected / at risk) | 17/109 | 14/110 | 12/86
Other Adverse Events (participants affected / at risk) | 88/109 | 84/110 | 60/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Gain Prevention (Group 1) (N=109) | Weight Loss Intervention (Group 2) (N=110) | Self-guided Intervention (Group 3) (N=86)
Severe distress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Heart Attack (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Low blood pressure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Asystole (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bloodstream Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Blockage in legs, stroke, surgery (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Clavicle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head Injury and amnesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Bleeding and ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ulcerative Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration and sinus infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Bladder Surgery (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Hysterectomy due to cervical cancer (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Knee Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Surgery for mass in large intestine (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cerebral Spinal Fluid leak and surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Biopsy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Heart Surgery (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0)
Back Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hip Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Foot Surgery (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1)
Prostate Surgery (cancer) (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Brain surgery (tumor) (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Gastric Sleeve Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hole in Heart (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Gain Prevention (Group 1) (N=109) | Weight Loss Intervention (Group 2) (N=110) | Self-guided Intervention (Group 3) (N=86)
Emotional Disturbance (Psychiatric disorders) | 6 (6) | 6 (6) | 0 (0)
Depression (Psychiatric disorders) | 27 (36) | 25 (33) | 29 (37)
High Blood Pressure (Cardiac disorders) | 18 (20) | 24 (25) | 11 (13)
Difficulty Sleeping (General disorders) | 18 (19) | 23 (25) | 25 (26)
Abnormal Dreams (General disorders) | 25 (25) | 15 (15) | 15 (17)
Rapid Weight loss (General disorders) | 0 (0) | 10 (11) | 0 (0)
Swelling (General disorders) | 7 (8) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 12 (13) | 15 (15) | 7 (8)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 9 (9) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 28 (32) | 25 (26) | 17 (17)
Constipation (Gastrointestinal disorders) | 6 (6) | 6 (6) | 5 (5)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0)
Cold (Infections and infestations) | 9 (12) | 15 (17) | 0 (0)
Influenza (Infections and infestations) | 7 (7) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT03156660/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03156660/SAP_001.pdf
  • Informed Consent Form (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT03156660/ICF_002.pdf